CLINICAL TRIAL: NCT07097311
Title: A Phase II, Open Label Study to Evaluate the Safety of Triheptanoin for the Prevention of Hypoglycemia in Patients With Medium Chain Acyl-CoA Dehydrogenase Deficiency (MCADD)
Brief Title: Study to Evaluate the Use of Triheptanoin in Patients With Medium Chain Acyl-CoA Dehydrogenase Deficiency (MCADD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jerry Vockley, MD, PhD (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Jerry Vockley, MD, PhD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25050173
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Medium-chain Acyl-CoA Dehydrogenase Deficiency
Keywords: Medium-chain Acyl-CoA Dehydrogenase Deficiency
MeSH Terms: conditions — Medium chain acyl CoA dehydrogenase deficiency | interventions — triheptanoin

STUDY DESIGN:
Intervention Model Description: The study will include 3 cohorts with up to 8 participants enrolled in each cohort. Cohort 1: ≥ 16 years of age; Cohort 2: 10-15 years of age; Cohort 3: 4-9 years of age. At least 2 participants will be enrolled in Cohort 1 to assess for any safety signals. If no safety issues are identified, enrollment in Cohort 2 will begin. At least 2 participants will be enrolled in Cohort 2 to assess for any safety signals before opening enrollment in Cohort 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1.0 gm/kg/day triheptanoin (Experimental): Up to 24 subjects (8: 4-9 years of age, 8: 10-15 years of age; 8: 16 years of age or older) will take 1.0 gm/kg/day divided into 3 or 4 doses
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Open-label design with doses of triheptanoin up to 1.0 gm/kg/day. The dose will be titrated from Day 1-24.
  Other Names: Dojolvi

SUMMARY:
This is a medical research study to test a medication in patients 4 years of age and older with a disease called medium-chain acyl-CoA dehydrogenase deficiency (MCADD). The medication is triheptanoin, which is currently FDA approved for the treatment of long chain fatty acid oxidation disorders (FAODs). Previous research suggests that triheptanoin may also be effective in the treatment MCADD. This study will investigate the safety and efficacy (how well it works) of triheptanoin patients with MCADD.

DETAILED DESCRIPTION:
Participation in the study will require four outpatient visits at the Clinical and Translational Research Center at the UPMC Children's Hospital of Pittsburgh (also called the PCTRC). The total length of the study participation is approximately 8 weeks.

Participants will come in for a screening visit (Visit 1) to where they will undergo some lab work testing to confirm they are eligible for the study. If it's determined that they are eligible, they will undergo training on the use of a continuous glucose monitor (CGM). They will be sent home and asked to wear the CGM for the next 10 days. This 10-day period is considered the run-in period.

Following the run-in period, participants will return to the site (Visit 2) in a fasting state. Fasting labs will be drawn, then the participant will be provided with a meal and they will then be dosed with triheptanoin. Following the dose of triheptanoin, the participant will be sent home with instructions on how to titrate (increase) the dose of triheptanoin over the next 28 days.

Following the 28 day dose titration period, the participant will return to the site (Visit 3) in a fasting state. Fasting labs will be drawn, then the participant will be provided with a meal and then will then be dosed with triheptanoin Following the dose of ACER-001, the participant will be sent home with continuous glucose monitoring and will be asked to log their triheptanoin doses as well as overnight fasting times.

Triheptanoin doses will be weight-based with the maximum dose being 1.0 gm/kg daily divided into 3 or 4 doses.

Participants will be asked to return approximately 2 weeks later for Visit 4 to complete the same procedures outlined for Visit 3.

Study staff will contact the participant by phone approximately 1 week after Visit 4 to follow up on any adverse events.

All study procedures will be done at no cost to the participants.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of MCADD with molecular confirmation
2. ≥4 years of age
3. Able to perform and comply with study activities placement of a continuous glucose monitor, IV catheter, and all blood draws.
4. Negative pregnancy test for all female subjects of childbearing age.
5. Signed informed consent by the subject or parent/guardian of minors.
6. All females of childbearing age and all sexually active males must agree to use an acceptable method of contraception throughout the study. Appropriate contraceptive methods include hormonal contraceptives (oral, injected, implanted, or transdermal), tubal ligation, intrauterine device, hysterectomy, vasectomy, or double barrier methods. Abstinence is an acceptable form of birth control, though appropriate contraception must be used if the subject becomes sexually active.
7. Willing and able to adhere to requirements for maintaining continuous glucose monitoring.

Exclusion Criteria:

1. Use of any investigational drug within 30 days of Screening (Visit 1).
2. Active infection (viral or bacterial) or any other intercurrent condition as reported by the subject or noted on physical exam at screening.
3. Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at increased risk by participating in this study.
4. Known hypersensitivity to triheptanoin
5. Breastfeeding or lactating females.
6. Subjects with type 1 or type 2 diabetes, or who take medications as part of their routine care that can cause hypoglycemia
7. Subjects who are taking medications in the antimetabolite drug class (e.g., hydroxyurea, 5-fluorouracil (5-FU), methotrexate) will be excluded; these medications can interfere with the DEXCOM sensor and cause inaccurate glucose readings

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE v5.0 | 8 weeks

SECONDARY OUTCOMES:
Length of time before glucose falls below 60 mg/dL | 8 weeks
  Comparison of the length of time each participant's glucose level stays above 60 mg/dL, comparing their values from the run-in period to the results obtained between Visits 3 and 4
Length of time before glucose falls below 70 mg/dL | 8 weeks
  Comparison of the length of time each participant's glucose level stays above 70 mg/dL, comparing their values from the run-in period to the results obtained between Visits 3 and 4

OTHER OUTCOMES:
Length of time before glucose falls below 80 mg/dL | 8 weeks
  Comparison of the length of time each participant's glucose level stays above 80 mg/dL, comparing their values from the run-in period to the results obtained between Visits 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Vockley, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No